CLINICAL TRIAL: NCT01207934
Title: Recombinant Human Leptin Therapy Effects on Insulin Action
Acronym: Leptin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Amgen (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 98-0643
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Type Two Diabetes Mellitus
Keywords: diabetes; obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Leptin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): saline placebo for fourteen days
  Interventions: Dietary Supplement: placebo
- low-dose leptin (Experimental): 30mg per day of recombinant methionyl human (r-met hu) leptin for fourteen days
  Interventions: Drug: low-dose leptin
- high-dose leptin (Experimental): 80mg per day of recombinant methionyl human (r-met hu) leptin for fourteen days
  Interventions: Drug: high-dose leptin

INTERVENTIONS:
Dietary Supplement: placebo — saline placebo
  Arms: placebo
Drug: low-dose leptin — 30mg per day of recombinant methionyl human (r-met hu) leptin for fourteen days
  Arms: low-dose leptin
Drug: high-dose leptin — 80mg per day of recombinant methionyl human (r-met hu) leptin for fourteen days
  Arms: high-dose leptin

SUMMARY:
Leptin therapy improves insulin sensitivity in people with leptin-deficiency but it is not known whether it improves insulin action in persons who are not leptin deficient. The purpose of the present study was to determine whether leptin therapy has effects on insulin action in obese subjects with type 2 diabetes mellitus (T2DM). A randomized, placebo controlled trial was conducted in obese subjects with newly-diagnosed T2DM. Subjects were randomized to treatment with placebo, low-dose, or high-dose leptin. Insulin sensitivity was measured.

DETAILED DESCRIPTION:
Leptin therapy improves insulin sensitivity in people with leptin-deficiency but it is not known whether it improves insulin action in persons who are not leptin deficient. The purpose of the present study was to determine whether leptin therapy has weight loss-independent effects on insulin action in obese subjects with type 2 diabetes mellitus (T2DM). A randomized, placebo controlled trial was conducted in obese subjects with newly-diagnosed T2DM. Subjects were randomized to treatment with placebo (saline), low-dose (30 mg/d), or high-dose (80 mg/d) recombinant methionyl human (r-met hu) leptin for 14 days. Multi-organ insulin sensitivity before and after treatment was evaluated by using the hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotopically labelled tracer infusions to measure glucose, glycerol and fatty acid kinetics.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes for less than ten years
* Body mass index 25 - 40
* hemoglobin A1C 7.5% - 12.0%
* fasting blood glucose between 90 and 240mg/dL

Exclusion Criteria:

* smoking
* pregnancy
* diabetes medications
* regular exercise (more than 3 hours per week)
* uncontrolled hypertension: systolic blood pressure greater than 160 or diastolic blood pressure greater than 95

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1998-08; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Mittendorfer B, Horowitz JF, DePaoli AM, McCamish MA, Patterson BW, Klein S. Recombinant human leptin treatment does not improve insulin action in obese subjects with type 2 diabetes. Diabetes. 2011 May;60(5):1474-7. doi: 10.2337/db10-1302. Epub 2011 Mar 16. PMID 21411512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from August 1998 to August 1999. All subjects were recruited via the Volunteer for Health system at Washington University School of Medicine.
Period: Overall Study
Arm/Group | Placebo | Low-dose Leptin | High-dose Leptin
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low-dose Leptin | High-dose Leptin | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (1.2) | 53 (2.9) | 54 (1.6) | 56 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9
  Male | 4 | 2 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Baseline Glucose Disposal - a Measure of the Body's Ability to Process Sugars.
Description: pre-treatment glucose disposal. In general, a high glucose disposal rate is a marker of healthy metabolic function. Glucose disposal is measured by tracking the amount of tagged glucose in the bloodstream over time. It is adjusted to subject body weight.
Time Frame: baseline
Measure: Mean (Standard Error); unit: mmol/kg body weight/minute
Groups:
- Placebo: 14 days on placebo (saline)
- Low Dose Leptin: 30mg leptin daily for fourteen days
- High Dose Leptin: 80mg leptin daily for fourteen days
Arm/Group | Placebo | Low Dose Leptin | High Dose Leptin
Number analyzed (Participants) | 6 | 6 | 6
mmol/kg body weight/minute | 14.3 (3.1) | 18.4 (3.6) | 16.7 (2.4)

2. Secondary Outcome: Baseline Plasma Leptin Concentrations
Description: Leptin is an endogenous hormone. Here we measure the pre-treatment concentration of naturally-occurring leptin in the blood.
Time Frame: baseline
Measure: Mean (Standard Error); unit: Micrograms/Liter
Arm/Group | Placebo | Low Dose Leptin | High Dose Leptin
Number analyzed (Participants) | 6 | 6 | 6
Micrograms/Liter | 27 (7) | 24 (8) | 35 (10)

3. Primary Outcome: Post-treatment Glucose Disposal. I.e. Glucose Disposal After Treatment With Leptin or Placebo.
Description: This is a measure of the body's ability to metabolize sugar after treatment with either leptin or a placebo. We compare the effect of leptin therapy on insulin-mediated stimulation of glucose disposal with that of placebo. In general, a high glucose disposal rate is a marker of healthy metabolic function. Glucose disposal is measured by tracking the amount of tagged glucose in the bloodstream over time. It is adjusted to subject body weight.
Time Frame: fourteen days
Measure: Mean (Standard Error); unit: mmol/kg body weight/minute
Arm/Group | Placebo | Low Dose Leptin | High Dose Leptin
Number analyzed (Participants) | 6 | 6 | 6
mmol/kg body weight/minute | 17.5 (2.5) | 20.7 (3.0) | 19.1 (3.3)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Leptin vs High Dose Leptin; The null hypothesis was that there would be no change in glucose disposal between the three groups (placebo, low dose leptin, and high dose leptin). Power calculations were done showing that 6 subjects in each arm was enough to detect a 35% between group difference in glucose disposal at the 0.05 level with 80% power; Test type: Superiority or Other; p > 0.05, ANOVA — ANOVA for reapeated measures was used to compare the three groups

4. Secondary Outcome: Post-treatment Plasma Leptin Levels
Description: plasma leptin levels after fourteen days ingestion of either leptin or placebo.
Time Frame: fourteen days
Measure: Mean (Standard Error); unit: Micrograms/Liter
Arm/Group | Placebo | Low Dose Leptin | High Dose Leptin
Number analyzed (Participants) | 6 | 6 | 6
Micrograms/Liter | 25 (5) | 76 (19) | 5024 (500)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Leptin; The null hypothesis is that treatment would not effect plasma leptin levels; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — a priori threshold for significance was set at p = 0.05; T-tests compared pre and post-treatment values
Statistical Analysis 2: Comparison: Placebo vs High Dose Leptin; null hypothesis was that plasma leptin levels would be equal after treatment in the placebo and high-dose leptin groups; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — a priori threshold for significance was p = 0.05

ADVERSE EVENTS:
Arm/Group | Placebo | Low-dose Leptin | High-dose Leptin
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes